CLINICAL TRIAL: NCT04902924
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Repeated Cold- and Warm Water Immersion on Performance Recovery
Brief Title: Cold and Warm Water for Performance Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Ron Clijsen, Head of research, University of Applied Sciences and Arts of Southern Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-00546
Record Dates: First submitted 2021-04-29; First posted 2021-05-26 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: cold water immersion; warm water immersion; muscle damage; recovery

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repeated cold-water immersion (Experimental): In this arm, the participants undergo repeated cold water immersion at 10°C for 2 x 5 min. Between the immersion, a break will be conducted 2.5 min. Participants will be immersed up to the iliac crest
  Interventions: Behavioral: repeated cold water therapy
- Repeated warm-water immersion (Active Comparator): In this arm, the participants undergo repeated warm water immersion at 40°C for 2 x 5 min. Between the immersion, a break will be conducted 2.5 min. Participants will be immersed up to the iliac crestParticipants will be immersed up to the iliac crest.
  Interventions: Behavioral: repeated warm water therapy
- Control (Other): In this arm, the participants undergo the control intervention which comprises to remain seated for 12.5 min. The participants, that will perform the muscle damaging protocol under hypoxia will also be treated with the control condition.
  Interventions: Other: control

INTERVENTIONS:
Behavioral: repeated cold water therapy — This information can be found the description of the experimental arm.
  Arms: Repeated cold-water immersion
Behavioral: repeated warm water therapy — This information can be found the description of the experimental arm.
  Arms: Repeated warm-water immersion
Other: control — This information can be found the description of the experimental arm.
  Arms: Control

SUMMARY:
The overall aim of this study is, to evaluate the effectiveness of repeated cold- and warm water immersion on performance recovery after muscle damage.

DETAILED DESCRIPTION:
Participants perform a muscle-damage protocol, which comprises 5x20 drop jumps. After the exercise protocol is finished, the participants will undergo one of three recovery interventions. Cold-water immersion, Warm-water immersion or the control-intervention. During the exercise protocol and the recovery intervention following parameters will be assessed: Blood oxygenation, Muscle oxygenation, heart-rate, skin temperature and core temperature.

Then, performance recovery will be assessed during the following 72 hrs (in a 24 hrs interval).

At each time-point, following measurements will be conducted: vertical-jump performance, maximum voluntary isometric contraction of the m.quadriceps femoris muscle, muscle swelling and delayed-onset of muscle soreness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* No surgeries
* No previous injuries
* Anticonceptiva allowed

Exclusion Criteria:

* Acute injuries or current pain situations
* Cryophobia
* Fear
* Pregnancy
* Raynaud syndrome
* Medication intake

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland
Locations (1):
- University of Applied Sciences and Arts of Southern Switzerland, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wellauer V, Clijsen R, Bianchi G, Riggi E, Hohenauer E. No acceleration of recovery from exercise-induced muscle damage after cold or hot water immersion in women: A randomised controlled trial. PLoS One. 2025 May 7;20(5):e0322416. doi: 10.1371/journal.pone.0322416. eCollection 2025. PMID 40333546
- [Derived] Hohenauer E, Bianchi G, Wellauer V, Taube W, Clijsen R. Acute physiological responses and muscle recovery in females: a randomised controlled trial of muscle damaging exercise in hypoxia. BMC Sports Sci Med Rehabil. 2024 Mar 22;16(1):70. doi: 10.1186/s13102-024-00861-1. PMID 38520001
- See also: Full-text of the publication — https://pmc.ncbi.nlm.nih.gov/articles/PMC12057877/pdf/pone.0322416.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (3.3) | 23.1 (3.6) | 23.1 (1.6) | 23.3 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Voluntary Isometric Contraction (N)
Description: maximun voluntary isometric contraction of the knee extensor muscle will be assessed.
Time Frame: baseline to 72 hours
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
Newton
  BL | 54.8 (14.9) | 65.8 (11.6) | 52.2 (14.1)
  24h | 33.8 (13.9) | 41.1 (11.4) | 29.3 (8.7)
  48h | 41.8 (16.4) | 47.9 (10.3) | 34.7 (12.3)
  72h | 45.0 (17.0) | 54.5 (11.8) | 40.4 (13.2)

2. Primary Outcome: Delayed Onset of Muscle Soreness (DOMS)
Description: delayed onset of muscle soreness will be measured using a 0-10 scale, where 0 indicated no soreness and 10 indicates maximum soreness of the knee extensor muscles
Time Frame: baseline to 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
units on a scale
  BL | 0.1 (0.1) | 0.1 (0.1) | 0.1 (0.1)
  24h | 6.3 (2.6) | 6.1 (2.5) | 6.3 (2.7)
  48h | 5.0 (2.8) | 5.9 (3.0) | 6.1 (3.1)
  72h | 2.9 (2.6) | 4.6 (3.1) | 3.3 (2.3)

3. Primary Outcome: Muscle Swelling
Description: swelling of the knee extensor muscle will be performed using a ultrasound device.
Time Frame: baseline to 72 hours
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
cm
  BL | 4.3 (0.5) | 4.8 (0.6) | 4.6 (0.5)
  24h | 4.6 (0.5) | 5.2 (0.6) | 4.8 (0.6)
  48h | 4.5 (0.5) | 5.1 (0.5) | 4.7 (0.6)
  72h | 4.4 (0.5) | 5.0 (0.6) | 4.6 (0.6)

4. Primary Outcome: Creatine-kinase (U/l)
Description: using a blood sample (6 ml), creatine-kinase will be assessed
Time Frame: baseline to 72 hours
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
U/l
  BL | 111.0 (41.5) | 214.3 (180.9) | 119.8 (50.2)
  24h | 573.5 (488.9) | 820.6 (517.7) | 455.0 (318.2)
  48h | 335.4 (256.9) | 441.2 (349.2) | 288.3 (200.9)
  72h | 205.9 (146.2) | 314.3 (321.8) | 191.4 (118.1)

5. Primary Outcome: Muscle Blood Oxygenation
Description: Muscle oxygenation saturation (SmO2) of the knee extensor muscle will be measured using near-infrared spectroscopy device. Oxygenated haemoglobin (oxyHb), deoxygenated haemoglobin (deoxyHb) and total haemoglobin (TotHb) were assessed in arbitrary units and SmO2 was calculated as oxyHb/TotHb x 100 value (%)
Time Frame: through recovery intervention up to 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of muscle oxygen saturation
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
percentage of muscle oxygen saturation
  BL | 68.7 (4.4) | 68.8 (3.8) | 70.0 (3.7)
  post exercise | 70.4 (7.7) | 71.1 (7.1) | 73.4 (5.9)
  post Intervention | 76.6 (5.8) | 76.6 (3.4) | 74.0 (4.8)
  10min | 73.6 (5.3) | 75.5 (5.1) | 75.0 (5.4)
  20min | 67.8 (2.7) | 74.7 (3.2) | 73.5 (6.6)
  30min | 64.4 (6.4) | 74.4 (3.9) | 73.0 (6.1)

6. Primary Outcome: Skin Temperature (°C)
Description: Skin temperature will be measured using a near infrared thermography camera
Time Frame: through recovery intervention up to 30 minutes
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
degree Celsius
  BL | 30.6 (0.9) | 31.2 (1.1) | 30.9 (0.9)
  post Exercise | 30.0 (0.9) | 29.9 (1.0) | 29.5 (1.7)
  post Intervention | 15.2 (2.5) | 35.2 (0.7) | 31.8 (1.0)
  10min | 24.8 (1.2) | 35.3 (0.5) | 32.3 (0.8)
  20min | 27.9 (1.1) | 34.9 (0.5) | 32.4 (0.8)
  30min | 29.2 (1.0) | 34.8 (0.7) | 32.5 (0.9)

7. Primary Outcome: Core Temperature (°C)
Description: core temperature will be measured using temperature pill that will provide real time values from the gastrointestinal region
Time Frame: through recovery intervention up to 30 minutes
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
Number analyzed (Participants) | 10 | 10 | 10
degree Celsius
  BL | 37.1 (0.4) | 37.1 (0.2) | 36.8 (0.4)
  post Exercise | 38.5 (0.2) | 38.4 (0.3) | 38.3 (0.2)
  post Intervention | 37.9 (0.2) | 38.5 (0.3) | 37.9 (0.3)
  10 min | 37.6 (0.2) | 37.8 (0.2) | 37.5 (0.2)
  20 min | 37.3 (0.2) | 37.5 (0.2) | 37.3 (0.2)
  30 min | 37.2 (0.2) | 37.5 (0.2) | 37.2 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the experiment (baseline) up to 72 hours.
Description: There was never a risk for a serious adverse event or all-cause mortality in the setup of this risk group A study.
Arm/Group | Repeated Cold-water Immersion | Repeated Warm-water Immersion | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04902924/Prot_SAP_000.pdf